CLINICAL TRIAL: NCT00006264
Title: A Phase II Trial Of Induction Therapy With Zidovudine, Interleukin-2, And Ganciclovir In The Treatment Of HIV Positive Primary Central Nervous System Lymphoma
Brief Title: Zidovudine Plus Interleukin-2 and Ganciclovir in Treating Patients With AIDS-Related Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: AMC-019; CDR0000068204 (Other: NCI)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma
Keywords: AIDS-related primary CNS lymphoma
MeSH Terms: conditions — Lymphoma | interventions — aldesleukin; Ganciclovir; Zidovudine

INTERVENTIONS:
Biological: aldesleukin
Drug: ganciclovir
Drug: zidovudine

SUMMARY:
RATIONALE: Antiviral drugs such as zidovudine and ganciclovir act against viruses and may be an effective treatment for HIV. Interleukin-2 may stimulate a person's white blood cells to kill lymphoma cells. Combining these treatments may be effective in treating AIDS-related primary central nervous system lymphoma.

PURPOSE: Phase II trial to study the effectiveness of combining zidovudine, ganciclovir, and interleukin-2 in treating patients who have AIDS-related primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of zidovudine, interleukin-2, and ganciclovir in patients with AIDS related primary central nervous system lymphoma.
* Determine the response rate and overall survival of these patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive zidovudine (AZT) IV and ganciclovir IV over 1 hour every 12 hours on days 1-14. Patients also receive interleukin-2 (IL-2) IV every 12 hours on days 1-14 and a combination antiretroviral therapy consisting of nucleoside reverse transcriptase inhibitors (one of which must be AZT), nonnucleoside reverse transcriptase inhibitors, and protease inhibitors. AZT and ganciclovir treatment continues for an additional 7 days if partial response is achieved.
* Maintenance therapy: Patients receive IL-2 subcutaneously 3 times a week for 6 months. Patients also receive oral ganciclovir 3 times a day and combination antiretroviral therapy (AZT allowed, but not required). Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 1 year, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 10-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV positive
* Diagnosis of central nervous system lymphoma by one of the following means:

  * Brain biopsy
  * Thallium spectroscopy scan in conjunction with CT scan or MRI after failing to improve with at least 2 weeks of antitoxoplasmosis therapy
  * Cerebral spinal fluid positive for Epstein Barr virus in conjunction with positive thallium spectroscopy scan
  * Thallium spectroscopy scan demonstrating a thallium retention index greater than 1
* Documented intracranial space occupying lesion
* No systemic non-Hodgkin's lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,000/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* Bilirubin and SGOT no greater than 3 times upper limit of normal
* No major hepatic dysfunction as evidenced by encephalopathy, ascites, or varices

Renal:

* Creatinine clearance at least 60 mL/min

Other:

* No prior other malignancy within the past 5 years except carcinoma in situ of the cervix, basal cell carcinoma of the skin, or Kaposi's sarcoma not requiring systemic therapy
* No active uncontrolled infection except HIV or Epstein Barr virus
* No known allergy to E. coli derived products
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2003-03 (Actual); Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Harrington, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Aboulafia DM, Ratner L, Miles SA, Harrington WJ Jr; AIDS Associated Malignancies Clinical Trials Consortium. Antiviral and immunomodulatory treatment for AIDS-related primary central nervous system lymphoma: AIDS Malignancies Consortium pilot study 019. Clin Lymphoma Myeloma. 2006 Mar;6(5):399-402. doi: 10.3816/clm.2006.n.017. PMID 16640817